CLINICAL TRIAL: NCT07132398
Title: The Efficacy of Slow - Tapering Versus Rapid - Tapering Glucocorticoid Strategies in Preventing Relapses of Neuromyelitis Optica Spectrum Disorder (NMOSD) When Combined With Inebilizumab: A Multicenter, Open - Label, Randomized Parallel - Controlled Clinical Trial
Brief Title: Slow vs. Rapid Glucocorticoids Tapering With Inebilizumab in NMOSD
Acronym: STARGlu-NMO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Chun-Sheng Yang, Clinical Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YG20250610
Record Dates: First submitted 2025-06-17; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Neuromyelitis Optica (NMO); Neuromyelitis Optica Spectrum Disorders (NMOSD)
Keywords: NMO; NMOSD; Inebilizumab; Glucocorticoids
MeSH Terms: conditions — Neuromyelitis Optica | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Slow-tapering glucocorticoids + Inebilizumab arm (Active Comparator)
  Interventions: Drug: Slow-tapering glucocorticoids + Inebilizumab
- Rapid-tapering glucocorticoids + Inebilizumab arm (Active Comparator)
  Interventions: Drug: Rapid-tapering glucocorticoids + Inebilizumab

INTERVENTIONS:
Drug: Slow-tapering glucocorticoids + Inebilizumab — Slow-tapering glucocorticoids+Inebilizumab arm: A 300 mg intravenous infusion of inebilizumab will be administered on Day 1 and Day 15, followed by 300 mg infusions every 26 weeks thereafter. Prednisone will be initiated at a daily dose of 60 mg as concomitant therapy with inebilizumab. The prednisone dose will be tapered as follows: a reduction of 5 mg every 2 weeks until reaching 20 mg/day(Week 16); thereafter, a reduction of 5 mg every 4 weeks until discontinuation (a total duration of 32 weeks for combined inebilizumab and glucocorticoids therapy).
  Arms: Slow-tapering glucocorticoids + Inebilizumab arm
Drug: Rapid-tapering glucocorticoids + Inebilizumab — Rapid-tapering glucocorticoids+Inebilizumab arm: A 300 mg intravenous infusion of inebilizumab will be administered on Day 1 and Day 15, followed by 300 mg infusions every 26 weeks thereafter. Prednisone will be initiated at a daily dose of 60 mg as concomitant therapy with inebilizumab, with a tapering schedule of 5 mg reduction per week until discontinuation (a total duration of 12 weeks for combined inebilizumab and glucocorticoids therapy).
  Arms: Rapid-tapering glucocorticoids + Inebilizumab arm

SUMMARY:
Neuromyelitis optica spectrum disorder (NMOSD) is a central nervous system autoimmune condition mainly involving the spinal cord, optic nerves, and area postrema. The anti-aquaporin-4 (AQP4)-Immunoglobulin G (IgG) is a specific biomarker for NMOSD. Glucocorticoids(GCs) are used as first-line treatment for NMOSD. Oral glucocorticoids tapering is always suggested following the pused therapy in the maintenance phase. Inebilizumab, a humanized monoclonal antibody targeting CD19, has been proven effective in preventing NMOSD relapses. This study aims to evaluate and compare the efficacy and differences between glucocorticoids slow-tapering and rapid-tapering strategies combined with inebilizumab in preventing relapses in AQP4-IgG-seropositive NMOSD patients following an acute attack, with the goal of determining the optimal approach to steroid tapering and discontinuation after initiation of inebilizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent and comply with the requirements of the study protocol.
2. Age ≥18 years, regardless of sex.
3. Diagnosis of NMOSD according to the 2015 International Panel for NMO Diagnosis (IPND) criteria.
4. Serum AQP4-IgG antibody positivity at screening.
5. An acute clinical attack (including the first attack) within 1 month before screening. After the acute attack was treated with high-dose corticosteroids, the current oral prednisone dose was reduced to 60 mg per day.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning to become pregnant during the study period.
2. Subjects with any serious acute, chronic, or recurrent infections (e.g., pneumonia, pyelonephritis, recurrent pneumonia, chronic bronchiectasis, tuberculosis, etc.).
3. Carriers of hepatitis B virus, or patients with chronic active hepatitis B or C, other chronic liver diseases, or HIV infection.
4. Abnormal liver function (ALT/AST >2 times the upper limit of normal); moderate to severe renal impairment (glomerular filtration rate <60 mL/min/1.73 m²).
5. Active malignancy.
6. Severe immunodeficiency.
7. Receipt of any B-cell depleting therapy within 6 months prior to initiation of baseline treatment, with B-cell counts below the lower limit of normal.
8. Receipt of other investigational treatments within 30 days prior to initiation of baseline treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
First adjudicated relapse event within 54 weeks | Baseline, 54 Weeks

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score from baseline at 54 weeks | Baseline, 54 Weeks
Change in Low-contrast Visual Acuity (LCVA) from baseline at 54 weeks | Baseline, 54 Weeks
Change in Timed 25-Foot Walk (T25-FW) test from baseline at 54 weeks | Baseline, 54 Weeks
Change in Expanded Disability Status Scale (EDSS) score from baseline at 106 weeks | Baseline, 106 Weeks
Change in Low-contrast Visual Acuity (LCVA) from baseline at 106 weeks | Baseline, 106 Weeks
Change in Timed 25-Foot Walk (T25-FW) test from baseline at 106 weeks | Baseline, 106 Weeks
Change in serum Neurofilament Light chain (sNfL) levels at 54 weeks | Baseline, 54 Weeks
Change in serum Glial Fibrillary Acidic Protein (sGFAP) levels at 54 weeks | Baseline, 54 Weeks
Change in serum AQP4-IgG titer at 54 weeks | Baseline, 54 Weeks
Change in serum Neurofilament Light chain (sNfL) levels at 106 weeks | Baseline, 106 Weeks
Change in serum Glial Fibrillary Acidic Protein (sGFAP) levels at 106 weeks | Baseline, 106 Weeks
Change in serum AQP4-IgG titer at 106 weeks | Baseline, 106 Weeks
Change in Visual Analogue Scale (VAS) score from baseline at 54 weeks | Baseline, 54 Weeks
Change in Visual Analogue Scale (VAS) score from baseline at 106 weeks | Baseline, 106 Weeks
Change in Quality of Life (QoL) score from baseline at 54 weeks | Baseline, 54 Weeks
Change in Quality of Life (QoL) score from baseline at 106 weeks | Baseline, 106 Weeks
Proportion of Relapse-free Participants at 54 weeks | Baseline, 54 Weeks
Proportion of Relapse-free Participants at 106 weeks | Baseline, 106 Weeks
Percentage of patients in glucocorticoid-free remission between 54 and 106 weeks | 54 Weeks, 106 Weeks
Annualized Relapse Rate (ARR) at 54 weeks | Baseline, 54 Weeks
Annualized Relapse Rate (ARR) at 106 weeks | Baseline, 106 Weeks
Daily and acumulate dose of glucocorticoids at relapse before 54 weeks | Baseline, 54 Weeks
Adverse events (AEs) and Serious AEs (SAEs) at 54 weeks | Baseline, 54 Weeks
Immunoglobulin levels at 54 weeks | Baseline, 54 Weeks
Pelvic X-ray at 54 weeks | Baseline, 54 Weeks
Adverse events (AEs) and Serious AEs (SAEs) at 106 weeks | Baseline, 106 Weeks
Immunoglobulin levels at 106 weeks | Baseline, 106 Weeks
Pelvic X-ray at 106 weeks | Baseline, 106 Weeks

OTHER OUTCOMES:
Lymphocyte Subpopulation Monitoring at 54 weeks | Baseline, 54 Weeks
Lymphocyte Subpopulation Monitoring at 106 weeks | Baseline, 106 Weeks

IPD SHARING:
Plan to Share IPD: No